CLINICAL TRIAL: NCT04986683
Title: Novel DWI Methods to Minimize Postoperative Deficits in Pediatric Epilepsy Surgery
Brief Title: Diffusion MRI Methods to Minimize Postoperative Deficits in Pediatric Epilepsy Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Justin Jeong-Won Jeong, Associate Professor, Wayne State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pediatric epilepsy DWI
Record Dates: First submitted 2021-07-22; First posted 2021-08-03 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Focal Epilepsy
MeSH Terms: conditions — Epilepsies, Partial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Patients with drug-resistant epilepsy (Experimental): All patients who undergo two-stage epilepsy surgery will receive two longitudinal evaluations of brain MRI and neuropsychology test: a month before surgery and 1.5 years after surgery.
  Interventions: Diagnostic Test: Brain magnetic resonance imaging; Behavioral: Neuro-psychology testing

INTERVENTIONS:
Diagnostic Test: Brain magnetic resonance imaging — Brain magnetic resonance imaging (MRI) will be done using multiple sequences to evaluate the presence, type, and severity of brain abnormalities in enrolled subjects.
  Other Names: MRI
Behavioral: Neuro-psychology testing — Participants will undergo age-appropriate neuro-psychology testing to assess motor, language, and other neurocognitive functions potentially affected by drug-resistant epilepsy.
  Other Names: neuro-cognitive testing; neuro-psychology

SUMMARY:
This project will test the accuracy of a novel diffusion-weighted magnetic resonance imaging (DWMRI) approach using a deep convolutional neural network (DCNN) to predict an optimal resection margin for pediatric epilepsy surgery objectively. Its primary goal is to minimize surgical risk probability (i.e., functional deficit) and maximize surgical benefit probability (i.e., seizure freedom) by precisely localizing eloquent white matter pathways in children and adolescents with drug-resistant focal epilepsy. This new imaging approach, which will acquire a DWMRI scan before pediatric epilepsy surgery in about 10 minutes without contrast administration (and also without sedation even in young children), can be readily applied to improve preoperative benefit-risk evaluation for pediatric epilepsy surgery in the future. The investigators will also study how the advanced DWMRI-DCNN connectome approach can detect complex signs of brain neuronal reorganization that help improve neurological and cognitive outcomes following pediatric epilepsy surgery. This new imaging approach could benefit targeted interventions in the future to minimize neurocognitive deficits in affected children. All enrolled subjects will undergo advanced brain MRI and neurocognitive evaluation to achieve these goals. The findings of this project will not guide any clinical decision-making or clinical intervention until the studied approach is thoroughly validated.

DETAILED DESCRIPTION:
This project will combine advanced brain MRI with detailed neuro-psychology evaluation, performed in children and adolescents affected by drug-resistant focal epilepsy, to address two main aims, each of them with the following research hypotheses:

AIM 1. To determine the accuracy of deep learning tractography-based benefit-risk analysis compared to a standard electrical stimulation mapping (ESM) which is the current clinical standard for detecting eloquent cortical regions before epilepsy surgery.

Hypothesis 1.1 In healthy controls, DCNN-based tract classification will localize eloquent cortices, which are significantly overlapped at both single shell DWI acquisition and generalized Q-sampling imaging, suggesting that the accuracy of this approach may not be significantly affected by the acquisition protocol.

Hypothesis 1.2 DCNN-based tract classification will achieve at least 93% accuracy for prospective detection of ESM-defined eloquent cortices, including patients with a high likelihood of functional reorganization.

Hypothesis 1.3 Preservation of DCNN-classified eloquent white matter pathways during surgery will predict the avoidance of postoperative deficits as accurately as the preservation of ESM-defined eloquent cortex.

Hypothesis 1.4 Preservation of surgical margins optimized by Kalman filter on retrospective data will achieve seizure control and avoidance of postoperative deficits in a prospective surgical patient cohort.

In this aim, the investigators will test the accuracy of a recently developed deep learning-based benefit-risk model, called deep convolutional neural network (DCNN) tract classification combined with Kalman filter analysis, for non-invasive detection of eloquent white matter pathways and optimization of surgical margin (i.e., the distance between epileptogenic area and eloquent area), resulting in seizure freedom and avoidance of functional deficits. Failure to identify eloquent areas in the proposed resection region can have potentially lifelong consequences, and overestimation or incorrect localization of the extent of the eloquent regions may lead to incomplete resection of the epileptogenic zone. Without optimizing the benefit-risk ratio, the minimum acceptable margin is highly variable across different settings, ranging from 0 to 2 cm across epilepsy surgery centers. The investigators will study whether the proposed benefit-risk model can standardize (or customize) epilepsy surgery of individual patients by accurately optimizing the margins of the eloquent white matter pathways to be preserved, which is ultimately essential to balance the benefit of seizure freedom with the risk of functional deficit. This proposed new imaging approach could change clinical practice for pediatric epilepsy surgery and is widely applicable for other types of neurosurgical procedures such as tumor resection.

AIM 2. To determine the accuracy of deep learning-based connectome analysis for prediction of long-term neurocognitive improvement following epilepsy surgery.

Hypothesis 2.1 Connectivity efficiencies preserved in specific modular networks of preoperative DCNN-based connectome, found to be associated with postoperative functional improvement on retrospective data, will accurately predict long-term functional improvement in a prospective patient cohort.

Hypothesis 2.2 Longer epilepsy duration will be significantly associated with more decreased efficiency in full-scale IQ modular network of preoperative DCNN-based connectome, thus suggesting that earlier surgery will yield better long-term full-scale IQ improvement.

Hypothesis 2.3 Patients with ipsilateral resections, who show signs of postoperative "crowding" (i.e., verbal IQ improvement at the expense of non-verbal function), will show decreased efficiency in non-verbal and increased efficiency in verbal IQ network of DCNN-based connectome in the contralateral hemisphere.

In this aim, the investigators will test if an advanced DWMRI approach integrating DCNN and connectome helps decide timely surgery by providing 1) preoperative imaging markers underlying high likelihood of postoperative neurocognitive improvements and 2) mechanistic insight in structural brain reorganization associated with postoperative verbal IQ improvement. A series of preoperative imaging markers called "local efficiency" that quantifies how efficiently neural connection is shared by neighboring regions will be evaluated at the levels of specific modular networks. We expect that these markers can identify long-term and specific neurocognitive consequences (and potential predictors of these) associated with surgical intervention and their neural correlates for specific neurocognitive functions. In addition, neuronal remodeling associated with a functional crowding effect, studied with DWMRI connectome improved by the DCNN tract classification, will provide a new mechanistic insight in compensatory processes for verbal IQ function in children and adolescents who undergo resective surgery to treat drug-resistant focal epilepsy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with drug-resistant focal epilepsy

   1. Age 3-19 years. 2. Planned two-stage epilepsy surgery with subdural electrodes.
2. Healthy control subjects 1. Age 5-19 years. 2. No cognitive, motor, and/or language impairment or clinical elevations on a measure of behavioral problems. 3. Brain MRI interpreted as normal.

Exclusion Criteria:

For all subjects:

1. History of prematurity or perinatal hypoxic-ischemic event. 2. Hemiplegia on preoperative neurological examination by pediatric neurologists. 3. Dysmorphic features suggestive of a clinical syndrome. 4. Diagnosis of any pervasive developmental or psychiatric condition which clearly predates the onset of seizures, including autism spectrum disorder, tic disorders, obsessive-compulsive disorder. 5. MRI abnormalities showing massive brain malformation and other extensive lesions that likely destroyed the contralateral tracts and severely affected i) spatial normalization accuracy in advanced normalization tools (ANTs), mutual information (MI) between native T1- MRI of Geodesic SyN transform and template T1-MRI < mean-3*standard deviation of MI in the healthy control group and ii) parcellation accuracy in surface-matching-based deformable registration, target registration error (TRE) of fine tetrahedra mesh between native T1- MRI brain surface and template T1-MRI brain surface > mean-3*standard deviation of TRE in the healthy control group. 6. History of claustrophobia. 7. Unsuccessful MRI showing head motion > 2 mm in DWMRI (i.e., voxel size of DWMRI) which is evaluated by NIH TORTOISE DWMRI motion artifact correction package. 8. Subject who cannot speak English.

Ages: 3 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of DCNN tract classification for detection of ESM-defined eloquent white matter pathways in healthy controls | During procedure
  Spatial overlap of DCNN tract classification (range: 0-100%, 0 indicating no overlap and 100% indicating complete overlap) will be evaluated between two different DWMRI scans of healthy controls: single-shell and generalized Q-sampling imaging (GQI) that are acquired on the same day. 14 ESM-defined eloquent pathways will be obtained using 14 DCNN tract classifications from the single-shell and GQI data, and the spatial overlap between single shell and GQI data (score: %) will be assessed per each pathway.
Accuracy of DCNN tract classification for detection of ESM-defined eloquent area that will be acquired a month after the DCNN tract classification in children with drug-resistant epilepsy | 1 month
  Spatial overlap (range: 0-100%, 0 indicating no overlap and 100% indicating complete overlap) will be measured between cortical terminals of DCNN-classified white matter pathways and their ground truth data: ESM-defined eloquent areas that will be acquired a month after the DCNN tract classification.
Accuracy of DCNN tract classification for prediction of eloquent white matter pathways providing no postoperative deficits that will be assessed at 1.5 years after surgery | 1.5 years
  Preservation (score: 1) vs. no preservation (score: 0) of preoperative DCNN-classified white matter pathways will be compared with presence (score: 1) vs. absence (score: 0) of postoperative deficits in primary motor, language, auditory, and visual functions that will be assessed at 1.5 years after surgery.
Accuracy of DCNN tract classification combined with Kalman analysis to predict optimal margin balancing maximal seizure freedom and minimal functional deficits that will be assessed at 1.5 years after surgery | 1.5 years
  Preservation (score: 1) vs. no preservation (score: 0) of preoperative DCNN-Kalman filter predicted surgical margin will be compared with presence (score: 1) vs. absence (score: 0) of postoperative deficits and seizure freedom that will be assessed at 1.5 years after surgery.
Strength of association between local efficiency of preoperative network and functional measure: full-scale IQ, verbal-IQ, non-verbal IQ, expressive language, receptive language, and motor function that will be assessed at 1.5 years after surgery | 1.5 years
  Local efficiency value (range: 0-1, 0 indicating no efficacy and 1 indicating the strongest efficacy) will be evaluated from full-scale IQ network, non-verbal IQ network, verbal IQ network, expressive language network, receptive language network, and motor network of preoperative DWMRI connectome data, respectively. Full-scale IQ (normal mean: 100, standard deviation: 15), verbal IQ (normal mean: 100, standard deviation: 15), non-verbal IQ (normal mean: 100, standard deviation: 15), expressive language score (normal mean: 50, standard deviation: 10), receptive language score (normal mean: 50, standard deviation: 10), and motor score (normal mean: 50, standard deviation: 10) will be also evaluated from neuro-psychology testing at 1.5 years after surgery. The correlation coefficient (range: 0-1, 0 indicating no correlation and 1 indicating complete correlation) will be evaluated between local efficiency and neuro-psychology score measured for each corresponding function.
Strength of association between local efficiency of preoperative full-scale IQ network and epilepsy duration that will be assessed at the time of preoperative MRI (Hypothesis 2.2) | Within 1 day
  Full-scale IQ (normal mean: 100, standard deviation: 15) will be assessed at the time of preoperative MRI scan. It will be associated with local efficiency (range: 0-1, 0 indicating no efficacy and 1 indicating the strongest efficacy) of preoperative full-scale IQ network and epilepsy duration (range: 0-19 years) that will be assessed within 1 day of preoperative MRI scan. The correlation coefficient (range: 0-1, 0 indicating no correlation and 1 indicating a perfect correlation) will be evaluated between full-scale IQ and local efficiency of preoperative full-scale IQ network.
Strength of association between local efficiency change of contralateral verbal-/non-verbal IQ network and verbal-/non-verbal IQ change that will be measured between 1 month before surgery and 1.5 years after surgery | 1.5 years
  Longitudinal change of local efficiency in contralateral verbal-/non-verbal IQ network (range: -1 - +1, -1 indicating a complete loss of local efficiency after surgery and +1 indicating a complete gain of local efficiency after surgery) will be measured from postoperative and preoperative DWMRI connectome data that will be measured between 1 month before surgery and 1.5 years after surgery, respectively. It will be then correlated with the longitudinal change of verbal/non-verbal IQ (range: -100 - +100, -100 indication a complete loss of verbal/non-verbal IQ after surgery and +100 indicating a complete improvement of verbal/non-verbal IQ after surgery) that will be measured between 1 month before surgery and 1.5 years after surgery. The correlation coefficient (range: 0-1, 0 indicating no correlation and 1 indicating a perfect correlation) will be calculated between two longitudinal changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne State University/Children's Hospital of Michigan, Detroit, Michigan, United States